CLINICAL TRIAL: NCT02849041
Title: Screening of Tobacco-induced Cancers by Low-dose CT-scanner and Identification of Circulating Tumor Cells
Acronym: DETeCTOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DETECToR
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Tobacco; Cancer; Screening; Psychology; Lung
Keywords: Circulating Tumor Cells; Lung
MeSH Terms: conditions — Neoplasms; Neoplastic Cells, Circulating | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening program (Experimental): Who consults or is hospitalized in a medical services or vascular surgery 'Paris Saint Joseph Hospital Group' (GHPSJ) or 'the European Hospital Georges Pompidou' (HEGP) for occlusive arterial disease or aneurysm the abdominal aorta. This population should accept to have a medical imaging Low-dose CT-scanner and an Identification of Circulating Tumor Cells on their blood. 30 first patients will be proposing to particpate to the psychologic sub-study by answering to a Psychological Questionnaires
  Interventions: Device: medical imaging; Biological: Identification of Circulating Tumor Cells; Procedure: Psychological Questionnaires

INTERVENTIONS:
Device: medical imaging — Low-dose CT-scanner
Biological: Identification of Circulating Tumor Cells — Research of circulating tumor cells in blood
Procedure: Psychological Questionnaires — The procedure of screening test could be stressful. "False positive" results can cause anxiety and lead to additional costs, as well as increased exposure to radiation and invasive medical examination. Although this is based on some objective results, there is a high probability of adverse psychological effects in case of false positives; so there is cause for concern in the short term anxiety associated with positive results and the use of additional tests during the intervals between screening phases. There is no data related to psychological distress potentially caused by the discovery of circulating tumor cells.

SUMMARY:
Tobacco smoke is the most common source of exposure to carcinogens in humans. Indeed, the smoke contains about 1010 particles per ml and 4800 chemical compounds, at least 66 are carcinogenic. Tobacco smoke is the leading preventable cause of cancer in humans since it is responsible for lung cancer, upper aerodigestive tract (mouth, pharynx, larynx, esophagus), nasal cavity and sinuses, stomach, pancreas, liver, bladder, kidney, uterine cervix, and some myeloid leukemias.

This study aims to evaluate the combined effect of the scanner and the search for circulating tumor cells (CTC) on screening for tobacco-related cancers, accompanying smokers to cessation and addressing the psychological impact this approach.

DETAILED DESCRIPTION:
Study Objectives:

The study takes two lines of research:

1 - Imaging and Research circulating tumor cells:

The main objective is to evaluate the diagnostic value of the couple scanner low intensity and speed search of circulating tumor cells (CTC-LDCT) for screening in a population at high risk of lung cancer.

The secondary objectives are:

1. / comparing the added diagnostic value of dual-CTC LDCT screening that screening with LDCT used alone as it was used in the NLST study for lung cancer screening;
2. / to assess the interest assess the diagnostic value of research of circulating tumor cells to identify extrapulmonary cancers associated with smoking; 3 / evaluate the psychological effects of screening (see psychological study).

2 - Psychological Study The main objective is to study the emotional and psychosocial consequences of LDCT screening in the specific context of circulating tumor cells. This is to identify 1 / specific mechanisms of fear, anxiety and mental distress, 2 / adaptation strategies that could be beneficial for other patients, 3 / specific stressors caused by the device screening and / or medical information given to patients.

The secondary objective is to adjust and improve the communication skills of health professionals in order to develop an appropriate framework to support the emotional and psychological aspects involved in the screening process when ( will be) used daily in clinical practice.

Study Design

1. - Imaging and Research circulating tumor cells This is a prospective cohort study, multicenter (hospitals attached to the University Paris Descartes), open, non-randomized, single arm. Each subject enrolled in the study will undergo three screening procedures. Patients with cancer prevalent in the first exam will be offered treatment after the balance sheet. Only subjects who do not have cancer at the first examination will return to the actual screening study in search of incident cases. The same sequence of evaluation will be repeated once a year for 2 years.
2. - Psychological Study To achieve the objectives, a qualitative study based on grounded theory ( "grounded theory") will be built. Grounded theory is a research methodology that studies the psychosocial processes to make them modeled theoretically. Since this method involves small samples of subjects, promotes flexibility of data collection and detailed analysis of the cases studied.

ELIGIBILITY:
Inclusion Criteria:

* Subject with at least a cumulative smoking 30 pack-years,
* Active or weaned smoking since less than 15 years,
* Who consults or is hospitalized in a medical services or vascular surgery 'Paris Saint Joseph Hospital Group' (GHPSJ) or 'the European Hospital Georges Pompidou' (HEGP) for occlusive arterial disease or aneurysm the abdominal aorta,
* Accepting the repeat CT scans and blood tests, as provided for by the protocol and additional investigations which might be necessitated by the detection of abnormality (s) to previous reviews,
* Accepting, in case of continuing active smoking, engage in smoking cessation process.

Exclusion Criteria:

* Bronchial history of cancer,
* Diagnosis and / or previous treatment of another cancer within 5 years prior to study entry, with the exception of skin tumors and non melanomatous carcinoma in situ,
* Anterior resection pulmonary parenchyma, severe respiratory failure against-indicating any invasive procedure on the lung,
* Signs of presence and / or symptoms that may be due to a pre-existing cancer (eg, unexplained weight loss of more than 10% of initial body weight over the last 12 months, hemoptysis, ...)
* ECOG activity index ≥ 2,
* Acute respiratory infection that led to antibiotic therapy within 12 weeks prior to study entry,
* Renal impairment does not authorize, where appropriate, a contrast agent injection,
* Comorbidity (s) may increase the risk of death during the course of the trial.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of the number of patients diagnosed by LDCT | Day 1, Month 6, Month 12
  number of patients diagnosed by LDCT (Low Dose CT-scanner)
Assessment change of the number of patients diagnosed with CTC identification | Day 1, Month 6, Month 12
  Number of patients diagnosed with CTC (Circulating Tumor Cells) identification

SECONDARY OUTCOMES:
Assessment of the psychologic impact of screening a cancer | Day 1,
  A psychologist-researcher attended with patient at the first consultation by the physician. The actual psychological study will be proposed as voluntary patients to participate (30 patients). It will consist of extensive interviews, lasting approximately 60 to 90 minutes, led by psychologist-researcher in principle without exceeding 3 interviews for each patient. These interviews will aim to assess the nature of the psychological impact that screening has had on you and your resources to cope

CONTACTS AND LOCATIONS:
Overall Officials: TREDANIEL Jean, PhD, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yannoutsos A, Fontaine M, Galloula A, Damotte D, Chatellier G, Paterlini-Brechot P, Meyer G, Pastre J, Duchatelle V, Marini V, Schwering KL, Lazareth I, Ghaffari P, Stansal A, Sanson H, Labrousse C, Beaussier H, Nasr NB, Zins M, Salmeron S, Messas E, Lajonchere JP, Emmerich J, Priollet P, Tredaniel J. Peripheral arterial disease and systematic detection of circulating tumor cells: rationale and design of the DETECTOR prospective cohort study. BMC Cardiovasc Disord. 2019 Sep 13;19(1):212. doi: 10.1186/s12872-019-1193-1. PMID 31519196